CLINICAL TRIAL: NCT00800995
Title: SOD as Antioxidant Treatment OF ARMD
Brief Title: Superoxide Dismutase (SOD) as Antioxidant Treatment OF Age Related Macular Degeneration (ARMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Pr Romanet, CHU Grenoble
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHUG-0501
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Age Related Macular Degeneration
Keywords: ARMD; SOD
MeSH Terms: conditions — Macular Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator)
  Interventions: Dietary Supplement: Sham
- SOD (Experimental)
  Interventions: Dietary Supplement: SOD

INTERVENTIONS:
Dietary Supplement: SOD
  Arms: SOD
Dietary Supplement: Sham
  Arms: Control

SUMMARY:
INTRODUCTION:

Acting directly on the anti-radical enzyme chain, the superoxide dismutase (SOD), a major enzyme of the anti-oxidant system, provides an alternative of the antioxidants treatment in ARMD. Its synthesis depends on the cellular oxygenated reactive species, and leads to the conversion of the superoxide ion (O2-) into hydrogen peroxide (H2O2). This compound is the cell watch guard continuously regulating a free radicals' detoxifying chain. Subsequently, by increasing the production of H2O2, the administration of SOD can trigger endogenous/internal antioxidant mechanisms.

Oral administration of SOD is possible in its galenic form, Glisodine. The purpose of this study was to evaluate the protective effect of SOD on the bilateralization of the disease.

ELIGIBILITY:
Inclusion Criteria:

* unilateral neo-vascular ARMD

Exclusion Criteria:

* other pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
difference on AREDS score, Month 24 - Month 0 | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Grenoble, Grenoble, France